CLINICAL TRIAL: NCT03022435
Title: Protective Mechanisms Against a Pandemic Respiratory Virus: B-cell, T-cell, and General Immune Response to Seasonal Influenza Vaccine. Year 4, 2012
Brief Title: T-cell And General Immune Response to Seasonal Influenza Vaccine (SLVP018) Year 4, 2012
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17219-2012; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: Inactivated influenza vaccine; Live, attenuated influenza vaccine; Adult and elderly identical twins; Adult fraternal twins
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group B: 18-30 yo identical twins (LAIV) (Other): Participants to receive FluMist® LAIV by nasal spray.
  Interventions: Biological: LAIV
- Group B: 18-30 yo identical twins (TIV) (Other): Participants to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group D: 40-64 yo identical twins (TIV) (Other): Participants to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group F: 65-100 yo identical twins (TIV) (Other): Participants to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group F: 65-100 yo identical twins (High-Dose TIV) (Other): Participants to receive High-Dose Fluzone® standard TIV
  Interventions: Biological: High-Dose TIV

INTERVENTIONS:
Biological: TIV — Influenza Virus Vaccine Suspension for Intramuscular Injection
  Other Names: Fluzone® standard TIV
  Arms: Group B: 18-30 yo identical twins (TIV); Group D: 40-64 yo identical twins (TIV); Group F: 65-100 yo identical twins (TIV)
Biological: High-Dose TIV — High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe
  Other Names: High-Dose Fluzone® TIV
  Arms: Group F: 65-100 yo identical twins (High-Dose TIV)
Biological: LAIV — Live, attenuated influenza vaccine for Intranasal Spray
  Other Names: FluMist®
  Arms: Group B: 18-30 yo identical twins (LAIV)

SUMMARY:
This study will investigate markers, mechanisms and define general predictors for immunological health by comparing influenza vaccine responses in monozygotic and dizygotic twins.

DETAILED DESCRIPTION:
The investigators plan to study the response to different influenza vaccines much more broadly and deeply across different age groups and with different vaccine modalities and to probe the influence of genetics on these responses using monozygotic and dizygotic twins. On an investigational basis, the investigators plan to compare various immunological responses, identify age-specific biomarkers or clusters of markers, quantify the frequency of influenza-specific T-cells pre- and post-vaccination, and determine the effective breadth of T-cell repertoire to an influenza vaccine within an individual as a function of age and to what degree this is genetically determined.

Twin group B will will be randomly assigned to receive a single dose of inactivated vaccine, either the trivalent inactivated influenza vaccine (TIV) or intranasal live, attenuated influenza vaccine (LAIV). Twin Groups C-E will receive a single administration of TIV. Group F, elderly participants, will be randomly assigned to receive a single dose of inactivated vaccine, either the standard dose or the high-dose TIV. Blood samples to conduct the assays described will be taken at pre-immunization, Days 7-10 and 28 post-immunization.

Groups A, C and E were not enrolled for this year of the five year annual study.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory adults, ages 18-30 years (identical or fraternal twin pairs), 40-64 years (identical or fraternal twin pairs) or 65-100 years (identical twin pairs).
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with trivalent inactivated influenza vaccine (TIV) or live attenuated influenza vaccine (LAIV) in Fall 2012
2. Allergy to egg or egg products, or to vaccine components (including gentamicin, gelatin, arginine or MSG (LAIV for Group B only), and thimerosal (if TIV multidose vials used)
3. Life-threatening reactions to previous influenza vaccinations
4. Active systemic or serious concurrent illness, including febrile illness the day of vaccination
5. History of immunodeficiency (including HIV infection)
6. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
7. Blood pressure >150 systolic or > 95 diastolic at Visit 1
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C
10. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays, topical steroids and inhaled steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
11. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
12. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
13. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
14. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except aspirin up to 325 mg.day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
15. Receipt of blood or blood products within the past 6 months or planned receipt of blood products prior to completion of study visits.
16. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
17. Receipt of inactivated vaccine 14 days prior to study vaccination, or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
18. Receipt of live, attenuated vaccine within 60 days of vaccination, or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
19. Need for allergy immunization (that cannot be postponed) during the study period V01 to V03 (~Day 28)
20. History of Guillain-Barre Syndrome
21. Pregnant or lactating woman
22. Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits.
23. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned blood donation prior to completion of Visit 03 ( ~28 Day after study vaccination)
24. A current member of the clinical study team.
25. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.
26. Asthma or history of wheezing (for Group B volunteers only)
27. Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV (for Group B volunteers only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University; Garry Nolan, PhD, Principal Investigator — Stanford University; Ann Arvin, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kay AW, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Holmes S, Blish CA. Enhanced natural killer-cell and T-cell responses to influenza A virus during pregnancy. Proc Natl Acad Sci U S A. 2014 Oct 7;111(40):14506-11. doi: 10.1073/pnas.1416569111. Epub 2014 Sep 22. PMID 25246558
- [Background] O'Gorman WE, Huang H, Wei YL, Davis KL, Leipold MD, Bendall SC, Kidd BA, Dekker CL, Maecker HT, Chien YH, Davis MM. The Split Virus Influenza Vaccine rapidly activates immune cells through Fcgamma receptors. Vaccine. 2014 Oct 14;32(45):5989-97. doi: 10.1016/j.vaccine.2014.07.115. Epub 2014 Sep 6. PMID 25203448
- [Background] Kay AW, Bayless NL, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Blish CA. Pregnancy Does Not Attenuate the Antibody or Plasmablast Response to Inactivated Influenza Vaccine. J Infect Dis. 2015 Sep 15;212(6):861-70. doi: 10.1093/infdis/jiv138. Epub 2015 Mar 4. PMID 25740957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Numbers listed in the tables reflect individual twins and not twin pairs.
Groups:
- Group D: 40 - 64 yo Identical Twins; Group F: 65-100 yo Identical Twins (TIV): Participants to receive Fluzone® standard TIV
Period: Overall Study
Arm/Group | Group B: 18-30 yo Identical Twins (LAIV) | Group B: 18-30 yo Identical Twins (TIV) | Group D: 40 - 64 yo Identical Twins | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-Dose TIV)
Started | 5 | 5 | 6 | 3 | 3
Completed | 5 | 5 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group D: 40 - 64 yo Identical Twins (TIV); Group F: 65 - 100 yo Identical Twins (TIV): Participants to receive Fluzone® standard TIV
- Group F: 65 - 100 yo Identical Twins (High-Dose TIV): Participants to receive High-Dose Fluzone® standard TIV
- Total: Total of all reporting groups
Arm/Group | Group B: 18-30 yo Identical Twins (LAIV) | Group B: 18-30 yo Identical Twins (TIV) | Group D: 40 - 64 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (High-Dose TIV) | Total
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.98 (4.26) | 22.98 (4.26) | 42.76 (1.93) | 73.45 (4.20) | 73.45 (4.20) | 42.14 (21.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 2 | 2 | 16
  Male | 1 | 1 | 2 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 2 | 2 | 6 | 3 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 6 | 3 | 3 | 16
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 6 | 3 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Group B: 18-30 yo Identical Twins (LAIV) | Group B: 18-30 yo Identical Twins (TIV) | Group D: 40 - 64 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (High-Dose TIV)
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3
Participants | 5 | 5 | 6 | 3 | 3

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Groups:
- Group F: 65 - 100 yo Identical Twins (High Dose TIV): Participants to receive High-Dose Fluzone® standardTIV
Arm/Group | Group B: 18-30 yo Identical Twins (LAIV) | Group B: 18-30 yo Identical Twins (TIV) | Group D: 40 - 64 yo Identical Twins | Group F: 65 - 100 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (High Dose TIV)
Number analyzed (Participants) | 5 | 5 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 28 of study participation
Description: Clinical assessment performed at each visit
Arm/Group | Group B: 18-30 yo Identical Twins (LAIV) | Group B: 18-30 yo Identical Twins (TIV) | Group D: 40 - 64 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (TIV) | Group F: 65 - 100 yo Identical Twins (High-Dose TIV)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No